CLINICAL TRIAL: NCT02751957
Title: Pilot Study to Improve Access to Early Intervention for Autism in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00064533
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Receives caregiver coaching version of the Early Start Denver Model (ESDM) intervention, delivered by non-specialist workers. ESDM is an evidence based, behavioral intervention for young children who have an autism spectrum disorder. It is a behavioral treatment informed by the principles of applied behavior analysis.
  Interventions: Behavioral: Early Start Denver Model

INTERVENTIONS:
Behavioral: Early Start Denver Model — The Early Start Denver Model is an evidence based, behavioral intervention for young children who have an autism spectrum disorder. It is a behavioral treatment informed by the principles of applied behavior analysis.

SUMMARY:
This Mentored Career Development Award will lay the foundation for a career focused on addressing two Grand Challenges in Global Mental Health priorities: 1) improving child access to evidence-based mental health care, and 2) reducing the duration of untreated illness by developing culturally-sensitive early interventions. The proposed research aims to assess implementation barriers and facilitators as well as the impact of a brief caregiver coaching early autism intervention adapted for use in a low resource setting. Data from this pilot study would inform scalable early autism intervention programs for implementation in underserved, low resource, and low-literacy populations globally.

DETAILED DESCRIPTION:
In this proposal, the investigator's aim is to adapt the caregiver coaching version of the Early Start Denver Model (P-ESDM) and conduct a pilot study to explore the impact of this adapted intervention on child and caregiver outcomes in an African setting as well as understand key facilitators and barriers to implementation of the intervention in this setting. Importantly, this work aligns with an objective of the Federal Interagency Autism Coordinating Committee Strategic Plan: to support community-based studies that assess the effectiveness of interventions in broader community settings including scalable early intervention programs for implementation in underserved, low-resource, and low-literacy populations. The Early Start Denver Model (ESDM) was the first empirically-validated comprehensive intervention for toddlers with Autism Spectrum Disorders (ASD). In a study of P-ESDM that parallels the proposed study, Vismara et al (2009) demonstrated that in a brief 12 week, 1 hour per week, P-ESDM program with parents of toddlers with ASD, all but one parent in the study acquired mastery of the ESDM techniques at or above the 85 percent criterion by the fifth to sixth intervention session as measured by the ESDM fidelity scale. Furthermore, high levels of correct implementation of the ESDM techniques were maintained at follow-up for those parents who met fidelity and completed the program, with average percent accuracy ranging from 93-97%. The brief intervention also resulted in sustained positive growth in child social communicative behaviors. More recently, in an NIH-funded randomized controlled trial (RCT), Rogers et al (2012) found that both P-ESDM and community interventions were associated with increases in language and cognitive outcomes and decrease in ASD symptoms, despite the fact that the community intervention involved a greater number of intervention hours. Specifically, a 10-point increase in verbal developmental quotient (DQ), a 4-5 point increase in overall DQ, and a decrease in social affect symptoms on the Autism Diagnostic Observational Schedule (ADOS) were found. Moreover, the intervention resulted in lower levels of parenting stress.

The site of the proposed study is the Center for Autism Research in Africa at the University of Cape Town (Director, Prof Petrus de Vries). South Africa offers a unique opportunity to study interactions among treatment, child, family, community and context, which act as facilitators or barriers of intervention implementation, thus providing preliminary information that could help match the right treatment to the right child and family. In a recent multisite P-ESDM RCT Estes and colleagues reported that that this parent coaching intervention helped to maintain parental adjustment directly after a child was diagnosed with ASD. However, the numbers of negative life events were a significant predictor of parenting stress and sense of competence. Child and caregiver factors, particularly prevalent in South Africa (eg. poverty, malnutrition, HIV/AIDS), are known to affect child cognitive and social-emotional development, as well as parenting stress. Gathering data on the feasibility and impact of a scalable early ASD intervention in an environment where other significant child and caregiver contextual challenges exist, offers a unique opportunity to examine broader contextual factors affecting intervention implementation. The investigator will therefore document the effects of broader contextual factors (for e.g. caregiver mental health, negative life events, HIV/AIDS, and poverty) on treatment impact. In addition, this study will further the understanding of how to implement mental health early interventions in a low and middle-income country (LMIC) context, by examining processes used to train and supervise non-specialist providers who will provide the caregiver coaching in this context.

The long term goal of this proposal is to advance understanding of affordable, sustainable early intervention strategies for developmental disorders, including ASD that would benefit all families regardless of resource availability.

Specific Aim #1: Adapt the P-ESDM treatment manual and training approach. P-ESDM is a brief, scalable caregiver-mediated early autism intervention.

Specific Aim #2: Pre-pilot the adapted P-ESDM training and intervention and refine methodological details of the experimental protocol. This will provide information on the structure, content, and feasibility of the adapted P-ESDM intervention and training approach.

Specific Aim #3: Pilot of the adapted P-ESDM with preschool aged children with ASD exploring the impact on: a) child social communication abilities and overall developmental outcome, and b) implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASD based on DSM-5 criteria by a developmental pediatrician.
* a caretaker who speaks isiXhosa, Afrikaans or English
* lives within an area served by the Red Cross Neurodevelopmental clinic;
* willing to participate in the intervention and be randomized to the intervention or control group.

Exclusion Criteria:

* a neurodevelopmental disorder of known genetic etiology (eg. Downs syndrome)
* significant sensory or motor impairment (e.g. cerebral palsy)
* major physical problems
* uncontrolled seizures
* IQ below 35 as measured by mean age equivalence score on the Griffiths Scales of Mental Development
* unable to attend 3 assessments and 12, 1-hour, weekly consecutive intervention sessions.

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
The Griffiths Scales of Mental Development: Change in developmental quotient and language subdomain developmental quotient | Baseline, 12 week, and 16 weeks
  The Griffiths Scales of Mental Development: a standardized developmental test for children birth to 96 months. The composite developmental quotient and the language subdomain developmental quotient will be used as outcome variables.
The Vineland Adaptive Behavior Scales: Changes in communication and socialization standard scores | Baseline, 12 week, and 16 weeks
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is an individually-administered measure of adaptive behavior that is widely used to assess individuals with intellectual, developmental, and other disabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Franz, MBChB, Principal Investigator — Duke University
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa